CLINICAL TRIAL: NCT05873972
Title: Multimodal Deep Learning Radiomic Nomogram for Evaluation of Response to Cetuximab in Patient With Colorectal Cancer Liver Metastasis
Brief Title: Multimodal Model for Efficacy Prediction Cetuximab in Colorectal Cancer Liver Metastasis Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC-MULTIMODAL-02 RESEARCH
Record Dates: First submitted 2023-02-17; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer Liver Metastases
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Active Comparator): Chemotherapy regimens are determined based on the clinical experience of specialists
  Interventions: Drug: Cetuximab
- ARM B (Experimental): Chemotherapy regimens are determined based on the multimodal deep learning signature
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — AEM A：The specialist's decision to add cetuximab to chemotherapy will be based on their own judgment
  ARM B：The patient's CT imaging,genetic mutation information were input into the signature, and the FOLFOX+cetuximab regimen was selected when the output label was 1. FOLFOX+bevacizumab chemotherapy regimen was selected when the output label was 0

SUMMARY:
Establishment and validation of the deep learning model of Cetuximab efficacy in simultaneous RAS wild unresectable CRLM patients

DETAILED DESCRIPTION:
Ras wild unresectable CRLM patients with primary tumor resection followed by Cetuximab in combination with chemotherapy were included in this study. The tumor response was assessed by local MDT group. Based on tumor response, almost 100 CRLM patients were classified into two groups (Clinician drived regimen vs Multi-omics model drived regimen). They will be the prospective cohort to validate our deep learning model for predicting Cetuximab efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Histologically proven colorectal adenocarcinoma;
3. Simultaneous liver-limited metastases;
4. Initially unresectable liver metastases determined by a local MDT;
5. Life expectancy of > 6 months;
6. RAS and BRAF V600E wild-type;
7. ECOG 0-1;
8. Available CT imaging before treatment.

Exclusion Criteria:

1. Previous systemic treatment for metastatic disease;
2. Previous surgery for metastatic disease;
3. Extrahepatic metastases;
4. Unresectable primary tumor;
5. Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation;
6. Acute or subacute intestinal obstruction;
7. Second primary malignancy within the past 5 years;
8. Drug or alcohol abuse;
9. No legal capacity or limited legal capacity;
10. Uncontrolled hypertension, or unsatisfactory blood pressure control with ≥3 antihypertensive drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 months
  response rate will be assessed by local MDT

SECONDARY OUTCOMES:
progression free survival | 3 years
  progression free survival will be assessed by local MDT every two months during treatment, and telephone follow-up every three month after treatment
overall survival | 3 years
  overall survival will be assessed by researchers every two months during treatment, and telephone follow-up every three month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan hosptial, Fudan University, Shanghai